CLINICAL TRIAL: NCT06780332
Title: A Phase 4 Study to Evaluate the Impact of a Rapid Drug Desensitization (RDD) Protocol for Adults with Phenylketonuria and Experiencing Hypersensitivity Reactions to Palynziq
Brief Title: Rapid Drug Desensitization Study in Adults Experiencing Hypersensitivity Reactions to Palynziq
Acronym: PALLADIUM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 165-402
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Phenylketonuria; PKU
Keywords: Phenylketonuria; PKU; Palynziq; pegvaliase
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- RDD (Experimental): Participants undergoing RDD to Palynziq
  Interventions: Drug: RDD to Palynziq

INTERVENTIONS:
Drug: RDD to Palynziq — Delivery of gradually increasing doses of Palynziq at fixed time intervals over the course of several hours to a cumulative dose equal to the reactive dose. Reactive dose is defined as the dose at which the reactive HSR occurred which led to treatment interruption or reduction of dose or dose frequency.

SUMMARY:
The purpose of this study is to determine if rapid drug desensitization (RDD) to Palynziq will improve drug tolerability and treatment persistence in adult patients on commercial Palynziq experiencing hypersensitivity reactions (HSRs) leading to treatment interruption or reduction of dose or dosing frequency. See Section 10.8 for full list of HSR preferred terms. Study details include:

* Study duration: Up to 30 weeks (up to 6 weeks for Screening, then RDD, and 24 weeks of follow-up)
* RDD duration: 1 day
* Palynziq dosing/follow-up duration: 24 weeks
* Palynziq dosing frequency: Individualized

DETAILED DESCRIPTION:
This is a Phase 4 study to evaluate the impact of RDD on adult (≥18 years old) participants with PKU who have experienced HSRs leading to treatment interruption or reduction of dose or dosing frequency while receiving commercial Palynziq. This is not a blinded study. All participants will undergo the same assessments: Screening, the RDD in clinic on Day 1, in clinic dosing on Day 2, followed by remote visits in weeks 2-24 post-RDD to monitor for HSRs and changes in Palynziq dosing. Remote visits will occur every other week from Week 2 through Week 12, then monthly until Week 24.

The total duration of participation in the trial will be approximately 30 weeks: up to 6 weeks for screening, followed by RDD and 24 weeks of post-RDD follow-up.

No Data Monitoring Committee (DMC) will be used for this trial.

ELIGIBILITY:
Inclusion Criteria:

* Age:

  1.Participants must be 18 years of age or older inclusive, at the time of signing the informed consent.
* Type of Participant and Disease Characteristics 2. Participants must have phenylketonuria and must have been receiving commercial Palynziq and enrolled in the REMS.

  3. Participants must have developed HSRs leading to treatment interruption or reduction of dose or dosing frequency (Graade 2 or above) while on Palynziq, and must be able to undergo RDD within 6weeks from the reactive HSR and last Palynziq dose.
* Sex and Contraceptive/Barrier Requirement 4. Males and females are eligible to participate in this clinical study. Contraceptive use is not required during the study. Please refer to the Pregnancy section of USPI for further information.
* Informed Consent 5. Participants must be capable of giving written informed consent as described in Section 10.1, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Medical Conditions:

  1. Participant may not have any kind of disorders that, in the opinion of the investigator, may compromise the ability of the participant to give written informed consent and/or comply with any aspect of the study, and/or where any aspect of participation would be medically inadvisable for the underlying disorder.
  2. Participant must not be pregnant on the day of the RDD.
  3. Participants with uncontrolled asthma, active upper repiratory infection or other active infections, or cardiovascular disease. Asthma control will be assessed using the Asthma Control Test at screening.
* Prior/Concomitant Therapies:

  4. Participants were not using antihistamine premedication(s) at the time of reactive HSRs.

  5. Participants are willing and able to resume and tolerate Palynziq at the reactive dose prior to the RDD.

  6. Participant must not be receiving concurrent injectables containing PEG with the exception of PEG-containing vaccines, such as COVID-19 vaccinations (see Section 6.7).

  7.Participants receiving beta blockers.
* Prior/Concurrent Clinical Study Experience 8. Participants may not be currently participating in an interventional study of any investigational product, device, or procedure, or any other BioMarin clinical trial or post-marketing study.

Other Exclusions 9. Participants must not be experiencing reactions that are not appropriate for RDD, including severe cutaneous adverse reactions (SCAR) as defined by the American Academy for Allergy, Asthma, and Immunology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
To determine if RDD to Palynziq improves drug tolerability and treatment persistence in adults with PKU experiencing HSRs leading to treatment interruption or reduction of dose or dosing frequency (reactive HSR). | 24 weeks
  Tolerance, defined as the ability to restart Palynziq at the dose at which the reactive HSR occurred (reactive dose) and escalate as appropriate within 24 weeks following the RDD, without requiring treatment interruption or reduction of dose or dosing frequency due to HSRs and reduction in occurrence of HSRs Grade 2 or above within 24 weeks following RDD

SECONDARY OUTCOMES:
To characterize the immune response to Palynziq following RDD | 24 weeks
  Change in PEG IgG and IgM, PAL IgG and PAL IgM, and C3/C4 from Baseline to after RDD and at Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (1):
- Uncommon Cures, Chevy Chase, Maryland, United States